CLINICAL TRIAL: NCT00500162
Title: Comparison of Two Tri-Luma® Maintenance Regimens in the Treatment of Melasma
Acronym: CLARA
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Galderma R&D (Industry)
Responsible Party: Gladerma, Galderma
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RD.03.SPR.29059
Record Dates: First submitted 2007-07-11; First posted 2007-07-12 (Estimated); Last update posted 2021-02-17 (Actual); Status verified 2009-03

CONDITIONS: Melasma
MeSH Terms: conditions — Melanosis

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator)
  Interventions: Behavioral: Tri-Luma Maintenance regimen
- 2 (Active Comparator)
  Interventions: Behavioral: Tri-Luma Maintenance regimen

INTERVENTIONS:
Behavioral: Tri-Luma Maintenance regimen

SUMMARY:
Melasma is an acquired, symmetric, irregular hypermelanosis on sun-exposed areas of the face, commonly seen in Latin American women. It is a very frequent disease, although its true incidence is unknown.

Melasma has historically been difficult to treat and therapy remains a challenge for this chronic condition.

Melasma being a relapsing disease, there is a real need to address how to maintain efficacy achieved after acute treatment. A previous 12-month trial has shown that Tri-Luma® applied once daily over a long-term period is safe and tolerable. However, there are no robust data available either on the efficacy of Tri-Luma® in long-term treatment or guidance for a maintenance dosage regimen with this product.

Investigations have been made through a feasibility work among Dermatologists from USA and Latin America to assess their current practice in terms of Maintenance Therapy. Two regimens appear to be prescribed frequently and will be compared in this study.

The expectation is that Tri-Luma® will be effective, in one of the two regimens explored, in maintaining the Melasma improvement achieved with a previous treatment of Tri-Luma®.

DETAILED DESCRIPTION:
This study will last 32 weeks (8 months) as a maximum. 11 visits will take place (Last visit of Initial Treatment Phase = Baseline of Maintenance Phase) Initial Treatment Phase : Visit 1 (Baseline), 2 (Week 2), 3 (Week 4), 4 (Week 6), 5 (Week 8), Maintenance Phase : Visit 1 (Baseline), 2 (Week 4), 3 (Week 8), 4 (Week 12), 5 (Week 16), 6 (Week 20) , 7 (Week 24)

ELIGIBILITY:
Inclusion Criteria:

* Subjects with a clinical diagnosis of moderate to severe Melasma
* Subjects with a Fitzpatrick skin type between I and V

Exclusion Criteria:

* Female subjects who are pregnant or planning a pregnancy during the study;
* Subjects with a wash-out period for topical treatments on the treated areas less than 2 weeks for corticosteroids, glycolic Acid (in daily care cream, Bleaching products, UV light therapy and sunbathing, Topical retinoids including retinol, and less than 3 months for Lasers, IPL, dermabrasion, peeling
* Subjects with a wash-out period for systemic treatments less than 1 month for Corticosteroids and hormone-replacement therapies (unless subjects have been on treatment for at least 3 months)
* Subjects who foresee intensive UV exposure during the study (mountain sports, UV radiation, sunbathing, etc...);

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 340 (Actual)
Dates: Start 2006-11; Primary Completion 2008-10 (Actual); Study Completion 2008-10 (Actual)

PRIMARY OUTCOMES:
Time to relapse during the Maintenance Phase

SECONDARY OUTCOMES:
Subject's Quality of Life questionnaire (MelasQol)at the end of each treatment phase/Early termination.

CONTACTS AND LOCATIONS:
Overall Officials: Karime HASSUN, MD, Principal Investigator — UNIFESP - Universidade Federal de São Paulo
Locations (2):
- UNIFESP - Universidade Federal de São Paulo, São Paulo, Brazil
- Hospital General de México - Servicio de Dermatología, Mexico City, Mexico